CLINICAL TRIAL: NCT07038837
Title: Cluster Randomised Non-inferiority Trial Comparing Malaria Incidence When Implementing R21/Matrix-M Synchronized With Seasonal Malaria Chemoprevention Distribution Versus R21/Matrix-M Given Routinely Through the EPI in Two Health Districts in Chad (CoSAV-R21)
Brief Title: Comparison of Two Strategies for Administering the R21-Matrix M Vaccine in a Context of Seasonal Malaria Transmission in Chad
Acronym: COSAV-R21
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Epicentre, Paris, France. (Unknown); Chad Ministry of Public Health Expanded Programme on Immunisation (EPI) (Unknown); Chad Ministry of Public Health National Malaria Control Programme (NMCP) (Unknown); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COSAV-R21
Record Dates: First submitted 2025-06-03; First posted 2025-06-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Malaria Infection; Malaria Vaccines
Keywords: Vaccine; Malaria; Implementation strategy; Children; CPS; Pediatric; synchronized; coverage; prevention; incidence; prevalence
MeSH Terms: conditions — Malaria | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Routine" arm (control) (No Intervention): primary series (3 doses) of R21/Matrix M administered throughout the year as part of the routine Expanded Programme on Immunisation (EPI), followed by a single booster six months after the 3rd dose.
- "Synchronised" arm (intervention) (Experimental): primary series (3 doses) of R21/MatrixM synchronized with a seasonal malaria chemoprevention (SMC) campaign, followed by a single booster 12 months after 1st dose was introduced.
  Interventions: Other: "Synchronised" arm (intervention)

INTERVENTIONS:
Other: "Synchronised" arm (intervention) — Vaccines received together with CPS
  Arms: "Synchronised" arm (intervention)

SUMMARY:
This is a two-arm, cluster-randomised, phase IV trial conducted in Chad to assess the protective efficacy and impact in real-life conditions of a new strategy for administering the R21/MM malaria vaccine, synchronized within a seasonal malaria chemoprevention (SMC) campaign, among children living in areas of high seasonal malaria transmission.

In this study, a cluster is defined as the catchment area of a primary care health centre. In Chad, each catchment area is known as a 'zone of responsibility' (French: Zone de Responsibilité' [ZR]).

Twenty-six (26) of the total 27 ZRs in the districts of Moïssala and Dembo will be randomized in a 1:1 ratio to receive a 4-dose (3 primary doses + 1 booster) R21/MM schedule either (1) integrated into the routine EPI vaccination program (the "Routine" control arm), or (2) synchronized with an annual seasonal malaria chemoprevention (SMC) campaign (the "Synchronized" intervention arm).

Malaria incidence: R21/MM effectiveness will be assessed using the incidence of biologically confirmed clinical malaria (trial primary endpoint). The incidence of clinical malaria will be determined through enhanced surveillance of malaria cases in health centres and hospitals over a 17-month period (August 2025 - December 2026).

Coverage surveys: Cross-sectional surveys (cluster sampling) will be carried out to measure R21/MM vaccine coverage, SMC coverage, coverage of other malaria prevention measures, and coverage of other EPI vaccines.

Nested case-control study: A sub-sample of children admitted to Moïssala District Hospital with severe clinical malaria will be offered the opportunity to participate in a nested case-control study designed to estimate the individual protective efficacy of R21/MM against severe malaria.

ELIGIBILITY:
Inclusion Criteria:

* • Routine arm

  1. Aged 6 to 11 months at the time of the first R21/MM vaccination (dose 1).
  2. Residing in a village participating in the study and randomized to the routine arm.
  3. Oral consent provided by the child's parent/guardian.

     * Synchronised arm

  <!-- -->

  1. Aged 6 to 59 months at the time of the first R21/MM vaccination (dose 1) during the first 3 rounds of SMC (2025).
  2. Residing in a village participating in the study and randomized to the synchronized arm.
  3. Oral consent provided by the child's parent/guardian.

Exclusion Criteria:

* Exclusion criteria for both arms according to Chad national EPI guidelines

Malaria vaccine is not recommended for children with known severe hypersensitivity:

* To a previous dose of a malaria vaccine
* To a previous dose of hepatitis B vaccine
* One of the components of the R21/MM vaccine

Mild illness - including respiratory tract infections, mild diarrhoea and fever below 38.5° C - is not a contraindication to R21/MM vaccination. Malnutrition and being HIV-seropositive are also not contraindications to R21/MM vaccination.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70000 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Malaria incidence in children who were aged 6-11 months when receiving their first dose R21/MM | From enrollment to Month 17 (Aug 2025- december 2026)
  To assess whether the R21/MM vaccine synchronized with SMC is non-inferior in preventing malaria (based on malaria incidence) compared to R21/MM administered as part of routine EPI in children who were aged 6-11 months when receiving their first dose R21

SECONDARY OUTCOMES:
Malaria incidence | from enrolment to Month 17 (Aug 2025- Dec 2026)
  Incidence of clinical malaria (biologically confirmed by RDT) in each study arm among children aged 6-59 months, irrespective of R21/MM vaccination status
R21/MM vaccination coverage | from enrolment to Month 17 (Aug 2025- Dec 2026)
  Proportion of children having received the appropriate number of doses for their age
Coverage of other malaria prevention measures | from enrolment to Month 17 (Aug 2025- Dec 2026)
  Proportion of children possessing, and proportion of children using, a long-lasting insecticidal net (LLIN) on the day before completing the coverage survey questionnaire
Coverage of other EPI antigens | from enrolment to Month 17 (Aug 2025- Dec 2026)
  o Proportion of age-eligible children vaccinated against measles-1 and measles-2.
Protective efficacy against severe malaria | From enrollment to Month 17 (Aug 2025- december 2026)
  Protective efficacy of vaccination with R21/MM will be measured at the individual level against severe malaria confirmed by RDT and microscopy. The protective efficacy will be calculated from the relative risk (RR) of developing severe malaria in vaccinated and unvaccinated children.
Proportional morbidity | From enrollment to Month 17 (Aug 2025- december 2026)
  o Proportion of all-cause morbidity registered at health centres attributed to uncomplicated malaria
R21/MM safety | From enrollment to Month 17 (Aug 2025- december 2026)
  o Frequency of reported serious adverse events (SAEs), adverse events following immunization (AEFI), Serious AEFIs and reported adverse events of special interest (AESIs) following R21/MM vaccination
Coverage of other malaria prevention measures | From enrolment to month 17 (Aug 2025- Dec 2026)
  SMC coverage: average number of doses received per child and proportion of children receiving 0 and 5 doses

CONTACTS AND LOCATIONS:
Locations (1):
- Medecin sans Frontières, Moïssala, Mandoul Region, Chad

IPD SHARING:
Plan to Share IPD: Undecided